CLINICAL TRIAL: NCT05666830
Title: A Study to Observe the Effect of One-step Application of Artificial Dermis on Burn and Plastic Wounds
Brief Title: One-step Application of Artificial Dermis
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-033
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants will be treated with artificial dermis that perfomed with STSG simultaneously.
  Interventions: Device: Lando® artificial dermal regeneration matrix

INTERVENTIONS:
Device: Lando® artificial dermal regeneration matrix — Participants will be treated with artificial dermis that perfomed with STSG simultaneously.

SUMMARY:
The goal of this observational study is to study the effectiveness of one-step application of Lando® artificial dermal regeneration matrix for burn and plastic wound repair.

The main question it aims to answer is: the effectiveness of one-step application of Lando® artificial dermal regeneration matrix, including the take rate of skin graft and the appearance recovery of the wound.

Participants will be treated with artificial dermis that perfomed with STSG simultaneously. According to the routine clinical practice, the take rate of split-thickness skin graft at about 2-3 weeks and the appearance recovery of the wound at 3 months and 6 months after the implantation were measured.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 70 years old.
2. Patients with non-infectious wounds of deep burns, full-thickness traumatic skin defects or plastic surgery that need to be repaired and reconstructed by artificial dermis.
3. Patients who voluntarily participate in this clinical trial and sign the informed consent form. When the subjects are under 18 years old or they have no capacity or limited capacity, they should have the consent and signature of the guardian or legal representative.

Exclusion Criteria:

1. Patients who need to participate in other clinical researchers within 30 days before or during the period of joining the group.
2. Patients with poor control of diabetes (those with fasting blood glucose ≥ 7.0mmol/L or glycosylated hemoglobin HbA1c ≥ 12% after drug control, transaminase > 1.5 times and other diabetic complications).
3. Other cases that researchers believe not suitable for the participants of the trial.

Max Age: 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-infectious wounds of deep burns, full-thickness traumatic skin defects or plastic surgery that require repair and reconstruction of dermal defects.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Take rate of skin graft | 2~3 weeks
  The percentage of the area of survival skin graft assessed by the Investigator.

SECONDARY OUTCOMES:
Effective rate of skin grafting | 2~3 weeks
  The rate that the number of cases with excellent or good result divided by the total cases participated.
  Excellent：take rate of skin graft>90%； Good：take rate of skin graft between 81% and 90%； Fair：take rate of skin graft between 61% and 80%； Poor：take rate of skin graft<60%。
Vancouver Scar Scale score of skin grafting site | 3 months
  Vancouver Scar Scale score of skin grafting site after 3 months assessed by the Investigator.
Vancouver Scar Scale score of skin grafting site | 6 months
  Vancouver Scar Scale score of skin grafting site after 6 months assessed by the Investigator.
Vancouver Scar Scale score of donor site | 3 months
  Vancouver Scar Scale score of donor site after 3 months assessed by the Investigator.
Vancouver Scar Scale score of donor site | 6 months
  Vancouver Scar Scale score of donor site after 6 months assessed by the Investigator.
Percentage of wound contraction | 3 months
  The Percentage that the area of skin grafting area divided by the original area.
Percentage of wound contraction | 6 months
  The Percentage that the area of skin grafting area divided by the original area.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
We are sorry to declaim that the individual participant data is in a state of confidentiality.